CLINICAL TRIAL: NCT03521141
Title: Developing Precision Smoking Treatment in the Southern Community Cohort Study
Brief Title: PRecision Interventions for SMoking in the SCCS
Acronym: PRISM-SCCS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Meharry Medical College (Other); Tennessee State University (Other)
Responsible Party: Principal Investigator, Hilary Tindle, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160331; 16-06-571 (Other: Meharry Medical College); HS2016-3815 (Other: Tennessee State University)
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco Use Cessation; Precision Medicine
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices; Nicotine Replacement Therapy; Varenicline

STUDY DESIGN:
Intervention Model Description: Assessing parallel precision care interventions (groups 1, 2) and control group.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to participant arm assignment until delivery of lab results at month 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Guideline-Based Care (GBC) (Other): GBC participants are 1) referred to the state quitline, 2) provided the NCI Clearing the Air smoking cessation program, and 3) asked to talk to their healthcare provider about potential lung cancer screening (LCS). Medication assignment is guided by standard guidelines and a conversation between the study tobacco counselor and the participant. Groups 1 and 2 also receive GBC counseling.
  Interventions: Drug: Nicotine patch; Drug: Varenicline; Behavioral: NCI "Clearing the Air"
- Nicotine Metabolite Ratio (PC-NMR) (Active Comparator): Group 1, nicotine metabolism. Medication is guided by nicotine metabolism.
  Interventions: Drug: Nicotine patch; Drug: Varenicline; Genetic: Nicotine metabolism; Behavioral: NCI "Clearing the Air"
- Respiragene (PC-Respiragene) (Active Comparator): Group 2, genetically-informed lung cancer risk score. Medication assignment is guided by standard guidelines and a conversation between the study nurse and the participant.
  Interventions: Drug: Nicotine patch; Drug: Varenicline; Genetic: Genetically-informed lung cancer risk score; Behavioral: NCI "Clearing the Air"

INTERVENTIONS:
Drug: Nicotine patch — FDA-approved smoking cessation pharmacotherapy
  Other Names: Nicotine Replacement Therapy
Drug: Varenicline — FDA-approved smoking cessation pharmacotherapy
  Other Names: Chantix
Genetic: Nicotine metabolism — Information on nicotine metabolism will be used to inform selection of medication.
  Arms: Nicotine Metabolite Ratio (PC-NMR)
Genetic: Genetically-informed lung cancer risk score — This intervention uses information from a person's genes and smoking and family medical histories to estimate lung cancer risk compared to current smokers.
  Arms: Respiragene (PC-Respiragene)
Behavioral: NCI "Clearing the Air" — A booklet-led intervention designed by the NCI to support cessation at any stage of a quitter's journey, whether they are still thinking about quitting, have made the decision to quit, or have already taken steps to quit and just need help maintaining their new lifestyle.

SUMMARY:
Precision Care (PC) interventions, developed with guidance from a Community Advisory Board (CAB), will be piloted in a Randomized Clinical Trial (RCT) of approximately 100 eligible, consenting daily smokers in the Southern Community Cohort Study (SCCS) who are willing to make a quit attempt with medication and who reside in TN or MS. Participants will be randomized 1:1:1 to 1 of 3 groups; (1) group one informs selection of medication with information on nicotine metabolism; (2) group two offers a genetically-informed lung cancer risk score, and (3) group 3 is Guideline-Based Care (GBC). All groups will be followed for 6 months. All RCT participants will receive FDA-approved smoking cessation medication, be referred to the shared TN/MS state quitline, and be offered the NCI "Clearing the Air" standard intervention. The primary outcome is feasibility of delivering the precision interventions in the SCCS population, as evidenced by ability to recruit, engage, and retain participants through end of study. Secondary outcomes, for which the study is not powered, will include risk perceptions, use of quit aids, lung cancer screening among those who are eligible, and smoking cessation.

DETAILED DESCRIPTION:
Cigarette smoking significantly increases the risk of cancer and improved cessation strategies are needed. Biologically-informed precision treatment could benefit smokers but is understudied.

Tennessee and Mississippi Smokers that responded to a previous survey indicating willingness to be contacted for a smoking cessation clinical trial will be assessed for eligibility via phone and, if eligible, provide verbal consent and administer a baseline survey. These participants will then mail in written consent, upon receipt of which their SCCS stored blood samples will be analyzed. During lab processing, a study tobacco counselor will call enrolled participants to assist with their quit plan and inform them of randomization status. Participants will complete telephone surveys at 1, 3, and 6 months. During the 6 month follow-up call, participants will also be given their previously-unreported lab results (i.e., information on nicotine metabolism or lung cancer risk). After receiving lab results, participants will complete a final brief questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Daily smoker of ≥5 cigarettes per day (CPD)
* Enrolled participant of the Southern Community Cohort Study (SCCS) who completed a prior survey indicating they were willing to be contacted regarding a smoking cessation clinical trial
* Residence in Tennessee (TN) or Mississippi (MS)
* Has stored blood sample with the SCCS
* Has established primary care provider (PCP)
* Medically eligible and willing to take varenicline and NRT

Exclusion Criteria:

* Currently taking medication to quit smoking
* enrolled, or planning to be enrolled, in another smoking cessation program
* Inability to give informed consent or participate due to cognitive disorder (e.g., dementia, severe intellectual disability)
* Unstable psychiatric illness (ER or hospitalized for psychiatric condition in past 6 months, change in psychiatric medications in past 3 months, or suicidal ideation in past 6 months)
* not able to send or receive mail
* no access to a telephone or inability to communicate by telephone
* unable to speak and read English
* history of seizures or Buerger's disease
* currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary A Tindle, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Maureen Sanderson, PhD, RD, MPH, Principal Investigator — Meharry Medical College; Rebecca Selove, PhD, MPH, Principal Investigator — Tennessee State University; William Blot, PhD, Principal Investigator — Southern Community Cohort Study, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers or institutions.

REFERENCES:
- [Derived] Lee SS, Senft Everson N, Sanderson M, Selove R, Blot WJ, King S, Gilliam K, Kundu S, Steinwandel M, Sternlieb SJ, Cai Q, Warren Andersen S, Friedman DL, Connors Kelly E, Fadden MK, Freiberg MS, Wells QS, Canedo J, Tyndale RF, Young RP, Hopkins RJ, Tindle HA. Feasibility of precision smoking treatment in a low-income community setting: results of a pilot randomized controlled trial in The Southern Community Cohort Study. Addict Sci Clin Pract. 2024 Mar 15;19(1):16. doi: 10.1186/s13722-024-00441-1. PMID 38491559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mailed and Phone outreach to enrolled SCCS participants.
Pre-assignment Details: Begin enrollment (Baseline survey) for verbal consent, randomize on receipt of written consent. Analysis performed on randomized participants who completed the Results Call (those who "began" the pilot trial).
Period: Overall Study
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
Started | 19 | 19 | 20
Completed | 18 | 19 | 19
Not Completed | 1 | 0 | 1
Not completed — Death | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants who completed the Results Call, allowing for the intervention to be assigned and begin
Groups:
- Total: Total of all reporting groups
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene) | Total
Number analyzed (Participants) | 19 | 19 | 20 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.49 [55.06 to 65.28] | 62.23 [58.54 to 65.32] | 57.92 [55.78 to 62.49] | 59.24 [56.09 to 64.92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 13 | 42
  Male | 4 | 5 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 19 | 20 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 14 | 17 | 47
  White | 3 | 5 | 2 | 10
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 20 | 58

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Ability to Retain Participants
Description: Feasibility of delivering precision care (PC) interventions in the Southern Community Cohort Study (SCCS), as evidenced by ability to recruit, engage, and retain participants through end of the study.
Time Frame: Full trial: Baseline - 6 month survey
Population: Randomized participants who completed the Results Call, allowing for the intervention to be assigned and begin
Measure: Count of Participants; unit: Participants
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
Number analyzed (Participants) | 19 | 19 | 20
Participants
  Started Pilot Trial (completed results call) | 19 | 19 | 20
  Still enrolled at end of pilot trial | 18 | 18 | 19
  Completed 6 month survey | 17 | 14 | 12

2. Secondary Outcome: Cessation History - Quit Attempts
Description: Participants who reported making a quit attempt during the trial, as defined by use of a quit aid or reporting "not at all" for current smoking at any timepoint
Time Frame: Full trial: Baseline - 6 month survey
Population: Randomized participants who completed the Results Call, and were enrolled in the study through the 6 month timepoint (i.e., not withdrawn nor deceased)
Measure: Count of Participants; unit: Participants
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
Number analyzed (Participants) | 18 | 19 | 19
Participants | 16 | 17 | 17

3. Secondary Outcome: Cessation History - Medication Use
Description: Participants who received, and those who subsequently used, a smoking cessation medication during the trial
Time Frame: Full trial: Baseline - 6 month survey
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
Number analyzed (Participants) | 18 | 19 | 19
Participants
  Received any cessation medication | 17 | 15 | 16
  Started/used any cessation medication | 14 | 9 | 14

4. Secondary Outcome: Cessation History - Quitline
Description: Participants who reported using the quitline ("phone support") at any point during the trial
Time Frame: Full trial: Baseline - 6 month survey
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
Number analyzed (Participants) | 18 | 19 | 19
Participants | 4 | 5 | 5

5. Secondary Outcome: Cessation History - Self-reported Abstinence
Description: Participants who self-reported abstinence at the 6 month survey
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
Number analyzed (Participants) | 18 | 19 | 19
Participants | 7 | 5 | 3

6. Secondary Outcome: Cessation History - Validated Abstinence
Description: Participants who completed a salivary cotinine sample; participants who biochemically-verified as abstinent (salivary cotinine ≤10ng/ml)
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
Number analyzed (Participants) | 18 | 19 | 19
Participants
  Salivary cotinine sample received by study staff | 5 | 3 | 3
  Validated as abstinent (cotinine ≤10ng/ml) | 3 | 2 | 2

ADVERSE EVENTS:
Time Frame: Full trial: Baseline - 6 month survey
Description: Assessed at each survey timepoint for randomized participants who completed the Results Call (those who "began" the pilot trial)
Arm/Group | Guideline-Based Care (GBC) | Nicotine Metabolite Ratio (PC-NMR) | Respiragene (PC-Respiragene)
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/19 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 19/19 | 18/19 | 17/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guideline-Based Care (GBC) (N=19) | Nicotine Metabolite Ratio (PC-NMR) (N=19) | Respiragene (PC-Respiragene) (N=20)
Agitation and/or Irritability (Psychiatric disorders) | 12 | 5 | 12
Anger (Psychiatric disorders) | 13 | 5 | 7
Depressed mood (Psychiatric disorders) | 11 | 9 | 8
Anxiety (includes nervousness and panic attacks) (Psychiatric disorders) | 8 | 7 | 7
Restlessness (General disorders) | 10 | 11 | 4
Abnormal dreams and/or nightmares (Nervous system disorders) | 6 | 3 | 7
Insomnia and/or other sleep (Nervous system disorders) | 12 | 12 | 9
Headaches (Nervous system disorders) | 11 | 8 | 5
Dizziness (General disorders) | 5 | 4 | 3
Nausea and/or vomiting (Gastrointestinal disorders) | 3 | 4 | 3
Fatigue (General disorders) | 8 | 8 | 6
Itching (Skin and subcutaneous tissue disorders) | 5 | 8 | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 10
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 5
Other symptom (General disorders) | 5 | 5 | 6
Hospitalization (Surgical and medical procedures) | 2 | 3 | 0 — Hospitalizations during the course of the study judged to be unrelated to study procedures

LIMITATIONS AND CAVEATS:
Due to the small sample size of this pilot feasibility study, we cannot draw conclusions about differences across study arms. Larger follow-up studies are needed to test the efficacy of these precision approaches compared to guideline based care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT03521141/Prot_SAP_001.pdf